CLINICAL TRIAL: NCT02520830
Title: Sustained Effects of Blueberry Polyphenols on Vascular Function in Healthy Individuals
Brief Title: Effects of Blueberry-polyphenols on Endothelial Function, Absorption and Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Dr. Ana Rodriguez Mateos, Heinrich-Heine University, Duesseldorf
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Blueberries
Record Dates: First submitted 2015-07-08; First posted 2015-08-13 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: blueberry polyphenols; Polyphenol metabolites; endothelial function; Molecular mechanisms of action; Vascular function; Healthy men

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blueberry Group (Active Comparator): Dietary Supplement: 22 gram freeze-dried blueberry powder per day
  Interventions: Dietary Supplement: Blueberry Group
- Placebo Group (Placebo Comparator): blueberry polyphenol deprived powder 22 gram per day
  Interventions: Dietary Supplement: Placebo Group

INTERVENTIONS:
Dietary Supplement: Blueberry Group — 22 grams freeze-dried blueberry powder per day. Sustained intake (2x 11 grams daily over 1 month) of a drink consisting on freeze-dried wild blueberry powder dissolved in water
  Arms: Blueberry Group
Dietary Supplement: Placebo Group — Sustained intake (2x 11 grams daily over 1 month) of a drink consisting in placebo powder dissolved in water
  Arms: Placebo Group

SUMMARY:
Diets rich in fruits and vegetables have been linked to favorable cardiovascular outcomes in epidemiological studies.

Dietary intervention studies with certain micronutrients have shown promising effects on surrogate parameters of vascular risk including blood pressure, endothelial function and cholesterol levels. Wild blueberries have gained attention due to their high content of phytochemicals and particularly anthocyanins. Whether wild blueberries can improve vascular function and health when given over relevant time periods and in relevant populations is not known. Therefore, it is the overall hypothesis of the study proposal that chronic consumption of wild blueberries can improve endothelial function, a prognostically validated surrogate of cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* healthy male subjects without clinical signs or symptoms of cardiovascular disease
* 18-70 years

Exclusion Criteria:

* cardiovascular disease
* acute inflammation
* cardiac arrhythmia
* renal failure
* heart failure (NYHA II-IV)
* diabetes mellitus
* C- reactive protein > 1mg/dl
* malignant disease

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Endothelial function | baseline and 1 month
  Determination of endothelial function by Flow mediated dilation (FMD) 0 and 2 hours postconsumption

SECONDARY OUTCOMES:
Pulse wave velocity | baseline and 1 month
  Measured by SphygmoCor 0 and 2 hours postconsumption
Blood pressure | baseline and 1 month
  automatical measurements, 0 and 2 hours postconsumption
Blood lipids | baseline and 1 month
  biochemical analysis, 0 and 2 hours postconsumption

OTHER OUTCOMES:
Plasma blueberry polyphenol metabolites | baseline and 1 month
  measured by liquid chromotography- mass spectrometry (LC/MS) 0 and 2 hours postconsumption
Peripheral blood mononuclear cell-derived gene expression analysis | baseline and 1 month
  exploratory measures; measured by Agilent Human GZ 4x44 v2 Microarray

CONTACTS AND LOCATIONS:
Overall Officials: Ana Rodriguez-Mateos, PhD, Principal Investigator — Division of Cardiology, Pulmonology and Vascular Medicine, University Hospital Duesseldorf; Christian Heiss, MD, Study Chair — Division of Cardiology, Pulmonology and Vascular Medicine, University Hospital Duesseldorf
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, University Hospital Duesseldorf, Düsseldorf, Germany

REFERENCES:
- [Derived] Rodriguez-Mateos A, Istas G, Boschek L, Feliciano RP, Mills CE, Boby C, Gomez-Alonso S, Milenkovic D, Heiss C. Circulating Anthocyanin Metabolites Mediate Vascular Benefits of Blueberries: Insights From Randomized Controlled Trials, Metabolomics, and Nutrigenomics. J Gerontol A Biol Sci Med Sci. 2019 Jun 18;74(7):967-976. doi: 10.1093/gerona/glz047. PMID 30772905